CLINICAL TRIAL: NCT00002989
Title: A Randomized Phase III Study to Assess Intensification of the Conditioning Regimen for Allogenic Stem Cell Transplantation (ALLO-SCT) for Leukemia or Myelodysplastic Syndrome With a High Risk of Relapse
Brief Title: Combination Chemotherapy With or Without Idarubicin and Peripheral Stem Cell Transplantation in Treating Patients With Leukemia or Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065526; EORTC-06962
Record Dates: First submitted 1999-11-01; First posted 2003-11-25 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-07

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; previously treated myelodysplastic syndromes; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Busulfan; Cyclophosphamide; Idarubicin; Melphalan; Radiotherapy

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: idarubicin
Drug: melphalan
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of idarubicin plus peripheral stem cell transplantation using the patient's own or donated stem cells in treating patients with leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the value of idarubicin added to the standard conditioning regimen of allogeneic and autologous stem cell transplantation in patients with leukemia or myelodysplastic syndrome at high risk of relapse. II. Determine time to recovery of polymorphonuclear neutrophil leukocyte (PMN) and platelet counts in these patients. III. Evaluate the rate and type of grade 3-4 toxicity, particularly mucositis, and the number of days with fever in these patients. IV. Determine the incidence of acute and chronic graft versus host disease (GVHD) in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease (acute myelogenous leukemia (AML) vs acute lymphocytic leukemia (ALL) or lymphoblastic leukemia (LL) vs myelodysplastic syndrome (MDS) or secondary AML vs chronic myelogenous leukemia (CML) vs non-Hodgkin's lymphoma vs multiple myeloma), stage of disease (if not CML, 1st complete response (CR) vs 2nd CR vs no 1st/2nd CR; if CML, 1st CR vs other phases), conditioning regimen (cyclophosphamide (CTX) and total body irradiation (TBI) vs busulfan (BU) and CTX vs other), source of donor (allogeneic vs autologous), T-cell depletion or autologous transplantation (no vs yes), and source of stem cells (bone marrow vs peripheral blood stem cell). Patients are randomized to receive a standard regimen or an intensified regimen. Standard pretransplant treatment: CTX on days -6 and -5 and TBI on days -4 through -2, or BU on days -8 through -5 and CTX on days -4 and -3, or BU on days -8 through -5 and melphalan IV on day -4. Intensified pretransplant regimens: I. Continuous infusion of idarubicin (IDA) over 48 hours on days -12 and -11, followed 5 days later with CTX on days -6 and -5 and TBI on days -4 to -2 II. IDA followed 5 days later with BU on days -8 through -5, and then CTX on days -4 and -3 III. IDA followed by BU on days -8 through -5 and melphalan IV on day -4. Stem cells are infused on day 0. Patients are followed every 3 months during the first 3 years, then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 207 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myelogenous leukemia (AML), acute lymphocytic leukemia (ALL), lymphocytic leukemia (LL) or myelodysplastic syndromes (MDS) with at least one of the following high risk criteria: T-cell depleted stem cells or autologous stem cells Second complete response (CR) Previous CNS involvement No CR First CR achieved more than 5 weeks after start of remission-induction therapy Poor prognostic cytogenetic features: t(9;22), t(8;14), t(11;14), 11q23 anomalies, -5/5q-anomalies, -7/7q-anomalies, +8, complex cytogenetics Postcytotoxic/secondary AML Chronic myelogenous leukemia (CML) with at least one of the following high risk criteria: T-cell depleted stem cells Not in first chronic phase Non-Hodgkin's lymphoma or multiple myeloma Autologous stem cells

PATIENT CHARACTERISTICS: Age: 16 to 60 Performance status: WHO 0-2 Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No severe heart failure requiring diuretics No ejection fraction of less than 50% Neurologic: No severe concurrent neurological or psychiatric disease Other: HIV negative No allogeneic stem cells from donors other than HLA identical sibling(s)

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 207 (Estimated)
Dates: Start 1997-03

CONTACTS AND LOCATIONS:
Overall Officials: Theo De Witte, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen
Locations (9):
- Institut Jules Bordet, Brussels (Bruxelles), Belgium
- France (3):
  - Hopital Edouard Herriot, Lyon
  - Hotel Dieu de Paris, Paris
  - Institut Gustave Roussy, Villejuif
- Eberhard Karls Universitaet, Tübingen, Germany
- Italy (2):
  - Ospedale San Eugenio, Rome
  - Azienda Policlinico Umberto Primo, Rome
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen